CLINICAL TRIAL: NCT01827345
Title: Effects of Vitamin D Supplementation on Fall Risk and Functional Outcomes in Older Adults With Insufficient Vitamin D Levels: A Pilot Study
Brief Title: Vitamin D as a Supplement Against Falls in Elderly Study
Acronym: D-SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-2013; 00085737-8 (Other: University of Florida)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Vitamin D Deficiency (10 ng/mL to 30 ng/mL)
Keywords: Vitamin D; Falls; Balance; Physical Function
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D (Experimental): Participants will take the Institute of Medicine's recommended daily dose of vitamin D (800 IU/day) for six months.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Participants will take the Institute of Medicine's recommended daily dose of vitamin D (800 IU/day) for six months.

SUMMARY:
The role of vitamin D deficiency on increased risk for falls and physical dysfunction is unclear. It is also unclear if taking vitamin D improves physical function and reduces fall risk in older adults. The purpose of this research study is to explore the effects of taking the recommended dose of vitamin D (800 IUs/day) for six months on fall risk and physical functional outcomes in older adults with low vitamin D levels. The investigators hypothesize that the participants will experience fewer falls and function better physically after taking vitamin D for six months.

DETAILED DESCRIPTION:
The role of vitamin D deficiency on increased risk for falls and physical dysfunction is unclear. It is also unclear if taking vitamin D improves physical function and reduces fall risk in older adults. This study will look at the potential effects of taking vitamin D regularly on falls and physical function in older adults. A total of 50 individuals with low vitamin D levels (i.e., serum 25-hydroxy Vitamin D range 10 ng/mL to 30 ng/mL) and a recent fall history will be enrolled into a six-month study. During the 6 months in this study, participants will receive capsules containing 800 IU vitamin D, in non-childproof bottles, for two 3-month periods. Participants will be asked to consume one capsule per day for the duration of this six-month study, as well as attend four study visits: Screening Visit, Baseline Visit, 3-Month Visit (in approximately 3 months from the baseline visit), and 6-Month Visit (in approximately 6 months from the baseline visit). During the screening visit, participants will fill out questionnaires, complete the mini-mental status exam, have their blood pressure and pulse taken, and a small sample of blood will be drawn from their vein. During the baseline visit, participants will fill out questionnaires, have their blood pressure, pulse, height, weight, and waist circumference taken, and perform several measures of physical function. Finally, a mouth swab will be performed and a staff member will collect a stool sample that you brought to the study visit. During the 3-Month Visit, participants will complete a questionnaire and have their blood pressure and pulse taken. During the 6-Month Visit, participants will repeat the questionnaires and measures that they performed during the Baseline Visit. The investigators hypothesize that the participants will experience fewer falls and function better physically after taking vitamin D for six months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Serum 25-hydroxy vitamin D >10 ng/mL and < 30 ng/mL
* Having had a fall at least twice in the past six months
* Provide informed consent

Exclusion Criteria:

* Failure to provide informed consent
* Self-reported myocardial infarction, cerebrovascular accident, or unstable angina within the past 6 months; New York Heart Association (NYHA) Class 3 or 4 congestive heart failure; aortic stenosis; chronic hepatitis; cirrhosis; kidney disease; solid organ transplantation; major psychiatric disorder; history of kidney stones or history of renal colic; history of nephrotic syndrome; history of primary hyperparathyroidism or renal tubular acidosis; history of hypercalcemia; cancer requiring treatment in the past three years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer);
* Other significant co-morbid disease (e.g. renal failure on hemodialysis) or severe psychiatric disorder (e.g. bipolar, schizophrenia) that would impair ability to participate in the exercise-based intervention
* Cognitive impairment (i.e., Mini Mental Status Exam score < 23) or history of significant head injury
* Current use of anabolic medications (i.e., growth hormones or testosterone), antidepressant medications, antipsychotic agents, monoamine oxidase inhibitors, anticholinesterase inhibitors (i.e., Aricept), anticoagulant therapies (aspirin use is permitted), or antibiotics for HIV or tuberculosis
* Dietary supplementation with > 800 IU/day of Vitamin D
* Hypercalcemia (calcium > 10.4 mg/dL), hypocalcemia (calcium < 8.6 mg/dL), or renal insufficiency (estimated glomerular filtration rate (GFR) < 50 ml/min)
* Serum aspartate (AST) or alanine transaminase (ATL) >3 times upper limit normal (UPN)
* High amounts of physical activity (i.e. running or bicycling) > 120 min/week
* Excessive alcohol use ( >14 drinks per wk )
* History of drug or alcohol abuse (i.e., more than 5 drinks/day for males or more than 4 drinks/day for females)
* Planning to leave the area in the next year
* Resting heart rate > 120 bpm
* Systolic blood pressure > 180 mmHg
* Diastolic blood pressure > 100 mmHg
* Vision or hearing impairment
* Participating in another clinical trial or has received an investigational product within 30 days prior to screening/enrollment

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of Falls | Change in 6 months
  Assess the change in number of falls participants have after taking vitamin D for six months.

SECONDARY OUTCOMES:
Six Minute Walk Test | Change in 6 Months
  Assess the change in gait speed on the Six Minute Walk Test after taking vitamin D for six months.
Short Physical Performance Battery (SPPB) | Change in 6 Months
  Assess the change in functional performance on the SPPB after taking vitamin D for six months.
Grip Strength | Change in 6 Months
  Assess the change in grip strength after taking vitamin D for six months.
Weight | Change in 6 Months
  Assess the change in weight after taking vitamin D for six months.
Waist Circumference | Change in 6 Months
  Assess the change in waist circumference after taking vitamin D for six months.
Perceived Level of Functioning as Measured by the Activity Measure for Post-Acute Care (AM-PAC) | Change in 6 Months
  Assess the change in perceived level of functioning as measured by the Activity Measure for Post-Acute Care (AM-PAC) after taking vitamin D for six months.
Medical Outcomes Study Short-Form Health Survey (SF-36) | Change in 6 Months
  Assess the change in health-related quality of life after taking vitamin D for six months.
Microbiome in the Human Colon | Change in 6 Months
  Assess the change in microbiome in the human colon after taking vitamin D for six months. Analyses of changes in bacterial diversity will be accomplished by deep sequencing of the ribosomal RNA, a highly conserved molecule that is used to classify bacteria.
Microbiome in the Human Mouth | Change in 6 Months
  Assess the change in microbiome in the human mouth after taking vitamin D for six months. Analyses of changes in bacterial diversity will be accomplished by deep sequencing of the ribosomal RNA, a highly conserved molecule that is used to classify bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Anton, PhD, Principal Investigator — University of Florida
Locations (1):
- Institute on Aging; University of Florida, Gainesville, Florida, United States